CLINICAL TRIAL: NCT01603043
Title: A Multicenter, Randomized, Single-Masked, Sham-Controlled, Proof-of-Concept Study of Intravitreal AL-78898A in Patients With Bilateral Geographic Atrophy (GA) Associated With Age-Related Macular Degeneration (AMD)
Brief Title: A Multicenter, Proof-Of-Concept Study Of Intravitreal AL-78898A In Patients With Geographic Atrophy (GA) Associated With Age-Related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-12-020
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Geographic Atrophy
Keywords: Geographic Atrophy; Age-Related Macular Degeneration; Intravitreal injection
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AL-78898A (Experimental): 1 intravitreal injection per month for up to 12 months
  Interventions: Drug: Al-78898A
- Sham Injection (Sham Comparator): 1 mock injection per month for 12 months
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Al-78898A — 0.400 milligrams (mg) per 50 microliters (μL) administered as an intravitreal injection
  Arms: AL-78898A
Drug: Sham injection — Mock injection administered as an empty hub without needle
  Arms: Sham Injection

SUMMARY:
The purpose of this study was to to demonstrate superiority of AL-78898A intravitreal (IVT) injections compared to sham injections by assessing mean geographic atrophy (GA) lesion size change from baseline at Month 12.

DETAILED DESCRIPTION:
Participants meeting inclusion/exclusion criteria were randomized in a 2:1 ratio to receive AL-78898A or a sham injection. The study eye was assessed before and after each injection to ensure that the injection procedure and/or study medication had not endangered the health of the eye. The Investigator determined each month whether the patient was eligible to receive the next injection. The study was terminated due to a high likelihood that continued enrollment would reach the predefined study stopping criteria based upon the number of patients with drug deposit formation, which made an assessment of efficacy futile.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent and comply with the protocol.
* Diagnosis of bilateral geographic atrophy (GA) of the macula secondary to age-related macular degeneration, confirmed within 14 days prior to randomization.
* Study eye: Maximum best-corrected visual acuity (BCVA) of 55 letters (20/80 Snellen equivalent) and a minimum BCVA of 20 letters (20/400 Snellen equivalent) at screening
* BCVA of 20 letters (20/400 Snellen equivalent) or better in the non treated eye at screening without conditions other than AMD that, in the opinion of the investigator, could cause a rapid loss of vision.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any history or current evidence of exudative ("wet") AMD in study eye.
* Retinal disease other than AMD in the study eye.
* Any ophthalmologic condition in study eye that reduces the clarity of the media and that, in the opinion of the Investigator interferes with ophthalmologic examination, such as advanced cataract or corneal abnormalities.
* Any ophthalmologic condition in study eye that prevents adequate imaging of the retina judged by the site or reading center.
* A history or current medical diagnosis of glaucoma or ocular hypertension in study eye.
* Any ophthalmic condition in study eye that may require surgery during the study period.
* Current ocular or periocular infection in the study eye.
* History of any disease or current use of medication expected to cause systemic or ocular immunosuppression, such as RESTASIS®.
* History of uveitis or endophthalmitis in the study eye.
* History of intraocular surgery (including cataract surgery) in the study eye within 90 days prior to dosing.
* History of intravitreal or periocular injection in the study eye at anytime.
* Participation in another interventional clinical study, or use of any experimental treatment for AMD or any other investigational new drug within 6 weeks or during active period of drug (whichever is longer) prior to the start of study treatment.
* History of any medical or psychiatric condition, or substance abuse, that in the Investigator's opinion is likely to interfere with the patient's participation in the study, or likely to cause serious adverse events during the study.
* Women of child bearing potential UNLESS they are using a highly effective method of birth control.
* Known or suspected allergy or hypersensitivity to fluorescein or other injectables.
* Other protocol-defined exclusion criteria may apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hosseini, MD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7 study centers located in the United States.
Period: Overall Study
Arm/Group | AL-78898A | Sham Injection
Started | 7 | 3
Completed | 0 | 0
Not Completed | 7 | 3
Not completed — Study Futility | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-78898A | Sham Injection | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in GA Lesion Size at Month 12 as Assessed With FAF Imaging
Description: Efficacy analysis was not conducted due to the termination of the study prior to the primary and secondary efficacy endpoints and the small number of enrolled patients.
Time Frame: Day 0 (injection visit), Month 12
Arm/Group | AL-78898A | Sham Injection
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Yearly GA Lesion Size Growth Rate
Description: as for outcome 1
Time Frame: Baseline (Day 0), up to Month 12
Arm/Group | AL-78898A | Sham Injection
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Change From Baseline in BCVA at Month 12
Description: as for outcome 1
Time Frame: Baseline (Day 0), Month 12
Arm/Group | AL-78898A | Sham Injection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (6 months). An Adverse Event (AE) was defined as any untoward medical occurrence in a patient administered a study treatment regardless of causal relationship.
Description: At each visit, after the patient had the opportunity to spontaneously mention any problems, the Investigator inquired about AEs by asking the standard questions, "Have you had any health problems since your last study visit?" and "Have there been any changes in the medicines you take since your last study visit?"
Arm/Group | AL-78898A | Sham Injection
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 4/7 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AL-78898A (N=7) | Sham Injection (N=3)
Conjunctival haemorrhage (Eye disorders) | 2 | 1
Eye pruritus (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Retinal oedema (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Product deposit (General disorders) | 4 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Dental implantation (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.